CLINICAL TRIAL: NCT05798585
Title: Comparing Erector Spinae Plane (ESP) and Thoracic Paravertebral (TPV) Block Analgesic Effect After Elective Video Assisted Thoracic Surgery (VATS): a Single Center, Randomized, Multiple-blinded, Controlled, Non Inferiority Trial
Brief Title: Comparing Erector Spinae Plane (ESP) and Thoracic Paravertebral (TPV) Block Analgesic Effect After Elective VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrea Saporito (Other)
Responsible Party: Sponsor-Investigator, Andrea Saporito, Head of Anesthesiology, PD DR MED, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TVPESP trial
Record Dates: First submitted 2023-01-13; First posted 2023-04-04 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Surgery; Thoracic

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- US-guided ESP block + sham US-guided TPV block (Experimental): ESP block will be performed with local anesthetic under US guide; instead TPV block with physiological solution
  Interventions: Procedure: ESP block
- sham US-guided ESP block + US-guided TPV block (Sham Comparator): ESP block will be performed with physiological solution under US guide; instead TPV block with local anesthetic
  Interventions: Procedure: ESP block

INTERVENTIONS:
Procedure: ESP block — US guided ESP infiltration (saline solution vs Ropivacaine 0.375% according to randomization): unilateral injection of 0,4 ml kg -1 (ideal weight)2 under US guidance between the deep fascia of erector spinae muscle and the two transverse processes at the level of the 5th thoracic vertebrae. Duration approximately 10-15 minutes

SUMMARY:
The aim of the study is to compare two different locoregional techniques in VATS.

DETAILED DESCRIPTION:
There are clear clinical and logistic reasons for pursuing the best possible post-operative pain management avoiding the negative side effects of opioid treatment; in order to garantee an enhanced recovery after surgery. A short hospital stay is fundamental to reduce patient morbidity and costs. Regional anesthetic nerve blocks are an ideal option to achieve this goal.

Paravertebral block serves as an ideal approach for thoracic and abdominal surgery through delivering segmental anesthesia of operative sites. Thoracic paravertebral block has superior analgesia as well as fewer complications than systemic opioids. It has been successfully applied in sternotomy, breast surgery, abdominoplasty, and laparoscopic cholecystectomy. ESP block is a recently described technique, with promising results in different scenarios. It probabily has a better risk profile than PVB, for its lower possibility of accidental pleural puncture and reabsorption of local anesthtetic than PVB one

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 year of age undergoing elective VATS lung resection at ORBV

Exclusion Criteria:

* patients with inability to consent, contraindications to standard care, or factors that can cause bias in interpretation, absolute contraindications to the regional anesthesia techniques studied (patient's refusal, allergy to local anesthetics, infections in the site of injection). Pregnant women are not a target study-group so they are excluded for design simplification. Conversion to the open technique will be a post-randomization exclusion factor concerning the main outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
cumulative dose of opioids at 24 and 48 h | 48 hours
  by using a PCA we will see how many times the patient asked for analgesia

SECONDARY OUTCOMES:
Pain scores at 4h, 8h, 24h, 48h via numeric rating scale (NRS) at rest and during cough | 48 hours
  we will test pain score in several moment by asking the NRS scale at rest and during cough
Hypotension | 48 hours
  we will compare the systolic pressure before anesthesia and after the block have been performed
Cardio-pulmonary complications | 48 hours
  we will check if any cardio-pulmonary complication is present after surgery during the hospital stay
Procedure time and complications | 48 hours
  we will observe the time necessary to perform the block and the complications after it
Need for anti-nausea medication (dosage, doses and time points) | 48 hours
  We will observe if the patient need any type of anti-nausea medication
Episodes of vomiting | 48 hours
  We will observe if any episode of vomiting is present
Episodes of urinary retention | 48 hours
  We will observe if any episode of urinary retention is present
Length of hospital stay | 48 hours
  We will observe how long the hospital stay is
Need for epidural catheter | 48 hours
  We will observe if the patient needs for an epidural catheter

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Saporito, Anesth, Study Chair — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Ente Ospedaliero Cantonale, Bellinzona, Bellinzona, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No